CLINICAL TRIAL: NCT01549483
Title: Differences in Small Airways Disease Between Asymptomatic and Symptomatic Subjects With Airway Hyperresponsiveness
Brief Title: Small Airways Disease in Asymptomatic and Symptomatic Subjects With Airway Hyperresponsiveness (AHR)
Acronym: ABHR
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, Dr., University Medical Center Groningen
Other Study IDs: ABHR001
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Asthma; Airway Hyperresponsiveness
Keywords: asthma; airway hyperresponsiveness; asymptomatic airway hyperresponsiveness; small airways
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal epithelium brushes for mRNA expression
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: asthmatic subjects
- Asymptomatic AHR: Asymptomatic subjects with airway hyperresponsiveness
- Control: Healthy controls, without airway hyperresponsiveness

SUMMARY:
The purpose of this study is to study differences in small airways (<2mm) parameters in asthma patients, subjects with asymptomatic airway hyperresponsiveness and healthy controls.

ELIGIBILITY:
Inclusion criteria for asymptomatic subjects with airway hyperresponsiveness (AHR) :

* Age between 18 and 65 years.
* Forced expiratory volume in one second (FEV1) > 80% predicted post bronchodilator.
* Provocative concentration causing a 205 fall in FEV1 (PC20) methacholine <8 mg/ml.
* No history of asthma or previous use of asthma medication.

Inclusion criteria for asymptomatic subjects without AHR :

* Age between 18 and 65 years.
* FEV1 > 80% predicted post bronchodilator.
* PC20 methacholine >8 mg/ml.
* No history of asthma or previous use of asthma medication.

Inclusion criteria for patients with asthma:

* Age between 18 and 65 years.
* FEV1 > 80% predicted.
* PC20 methacholine ≤8 mg/ml.
* Doctor's diagnosis of asthma.
* No history of Chronic obstructive pulmonary disease (COPD).

Exclusion Criteria:

* Use of inhaled or oral steroids, antihistamines, nedocromil, theophylline, leukotrien antagonists or long-acting beta-agonists for at least three weeks before the start of the study.
* Any disease that may affect the outcome of the study as judged by the Investigator.
* FEV1 <1.2 liter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out-patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Peripheral airway resistance measured with impulse oscillometry (IOS) | visit 1
  Difference between resistance at 5 Hz (R5) and resistance at 20 Hz (R20) (R5-20).

SECONDARY OUTCOMES:
Small airway parameters | visit 1
  Forced expiratory flow between 25 and 75% of forced vital capacity (FEF25-75), alveolar nitric oxide (NO), residual volume (RV), RV/total lung capacity (TLC)
mRNA expression in nasal epithelium | visit 2
Peripheral airway resistance measured during provocation test | visit 2
  Resistance at 5 Hz (R5) during a bronchial provocation test with methacholine

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Van den Berge, M.D., PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands